CLINICAL TRIAL: NCT04668859
Title: Midodrine as Novel Treatment of Post-Cardiopulmonary Bypass Vasoplegic Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI relocated
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-097
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Use of Midodrine in Post-cardiopulmonary Bypass Vasoplegic Syndrome
MeSH Terms: interventions — Midodrine; Methylcellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Midodrine Arm (Active Comparator): Patients will receive the drug Midodrine
  Interventions: Drug: Midodrine
- Placebo Arm (Placebo Comparator): Patients will receive placebo.
  Interventions: Drug: Methylcellulose

INTERVENTIONS:
Drug: Midodrine — Oral vasoactive that is metabolized by the liver an peripheral tissues into desglymidodrine, an active metabolite. It produces arteriolar and venous constriction with a subsequent elevation in blood pressure.
  Arms: Midodrine Arm
Drug: Methylcellulose — Placebo will consist of inert methylcellulose
  Arms: Placebo Arm

SUMMARY:
Vasoplegic syndrome (VS) is a common and serious complication of cardiopulmonary bypass (CPB) procedures associated with a significant increase in morbidity and mortality. VS is defined as significant hypotension, high or normal cardiac outputs, low systemic vascular resistance, low cardiac filling pressures, and vasopressor requirement despite adequate fluid resuscitation following CPB. Extensive research has been performed regarding the pathophysiologic response to CPB and risk factors associated with VS. No safe and effective preventive strategy has gained widespread use. Supportive care with intravenous (IV) vasopressors has thus been adopted as standard of care. The use of these medications, while effective in the majority of patients, generally necessitates close monitoring in an intensive care unit (ICU) setting. These patients are subject to prolonged ICU and hospital stays, as well as the potential complications of prolonged use of central venous lines (CVL) required to give these medications. Recent studies suggest midodrine, a generic oral vasopressor, may accelerate the decline in IV vasopressor requirements in select ICU patients. At our institution, the addition of midodrine to IV vasopressors for the treatment of VS has been observed to be effective in reducing IV vasopressor duration. No literature exists describing the use of midodrine in this patient population. The goal of this study is to investigate the novel use of midodrine in CPB surgery complicated by VS. Ultimately, we hope to produce literature supporting its use that may be applied on a global scale to improve patient care

ELIGIBILITY:
Inclusion Criteria:

* post-cardiopulmonary bypass surgery
* vasoplegic syndrome criteria

  1. MAP < 65mmHg
  2. Cardiac index>/=2.4 L/min/m^2, as determined by Swan-
  3. systemic vascular resistance index </=1400 dynes s/cm^5/m^2
  4. adequate fluid resuscitation as determined by treating critical care team
* vasopressor requirement

  1. norepinephrine 0.05-0.5 mcg/kg/min WITH/WITHOUT
  2. vasopressin any dose

Exclusion Criteria:

* allergy to midodrine
* pregnancy
* midodrine or cardiac glycoside as preadmission medication
* history of orthostatic hypotension, thyrotoxicosis, or pheochromocytoma
* severe organic heart disease (endocarditis, untreated congenital or rheumatic heart disease)
* liver failure/cirrhosis
* chronic kidney disease (GFR <30mL/hr)
* ventricular assist device implantation procedure, intra-aortic balloon pump placement, or heart transplantion
* unresolved post-operative acute kidney injury (rise in serum creatinine by >/= 0.5mg/dl from baseline
* inadequate tissue oxygenation (lactate > 2 mmol/L)
* inability to take oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Time from procedure end until discontinuation of IV vasopressors | 12 months

SECONDARY OUTCOMES:
Rate of decline in IV vasopressor dose | 12 months
Time until CVL removal | 12 mothns
ICU length of stay | 12 months
Hospital length of stay | 12 months
Rate of major infections/complications | 12 months
Rate of in-hospital and 30-day mortality | 12 months

IPD SHARING:
Plan to Share IPD: No